CLINICAL TRIAL: NCT05914493
Title: The Effect of Posture on Cognitive Function in Early Adolescence Athletes
Status: Completed | Type: Observational
Sponsor: Atılım University (Other)
Responsible Party: Principal Investigator, NAİME ULUG, PhD, Atılım University
Other Study IDs: E-59394181-604.01.02-62365
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Posture; Cognitive Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The effect of posture on cognitive function in early adolescence athletes — Posture evaluation:
  The form of Corbin et al. will be applied.
  Evaluation of cognitive functions:
  Basically, the Stroop test will be used, which evaluates the concentration and maintenance of attention depending on time and the task given.

SUMMARY:
While previous studies focused on the motor system in the analysis of postural functions, recently many researchers have determined that the sensory-cognitive-motor network system is required to determine the correctness of an action. , stroke individuals, Alzheimer's patients, Parkinson's disease, individuals with multiple sclerosis were discussed. In line with these studies, we can say that posture is handled with cognitive skills in people whose physical performance has decreased. However, the relationship between cognitive skills and posture in individuals with high physical performance has been ignored. Understanding posture and cognitive mechanisms is important both for physiotherapists who deal with posture from the neurophysiological aspect and for those who work in the field of psychology who deal with cognitive skills with its psychosocial aspect. The aim of the study is to reveal the relationship between posture and cognitive skills evaluated using the Stroop Test in healthy athletes in early adolescence.

DETAILED DESCRIPTION:
One of the important neuropsychological tests in evaluating cognitive performance is the Stroop Test. Basically, it evaluates the concentration and maintenance of attention depending on the time and the task given. It can also reveal the disruptive effects of perceptions on each other. The most interesting effect of the test is that it relates to changing the perception target or perceptual setup (set). It reveals the ease with which one's perceptual setup can be changed in line with changing demands and especially under a "disruptive influence", the ability to suppress a habitual behavior pattern and to engage in an unusual behavior. These are about flexibility and perceptual setup, attention and behavior shifting abilities. In cases where this ability is insufficient, perseverative, stereotypical, non-adaptive behaviors and difficulties in regulating and controlling motor movements occur. Accordingly, Stroop Test performance reflects the individual's degree of cognitive rigidity-flexibility. These functions are basically related to the frontal lobe activities of the brain. As a matter of fact, excessive impairments in such functions and in the ability to program behavior in general directly indicate a disorder in the frontal regions of the brain. It is stated that the Stroop test is also suitable for examining information-processing speed, automatic and parallel processing in cognitive processes. Indeed, the Stroop Test; It is a critical experimental task often used in the study of information processing speed and automatic and parallel processing models. When the literature is examined, the Stroop Test, which deals with the concept of 'mental flexibility', which is an important pillar of cognitive functions, is evaluated as a short-term standing or sitting posture only during the application of the test, while the possible effect of posture on cognitive functions was ignored by examining the normal postures of individuals. Revealing the relationship between posture and cognitive skills depending on brain areas is important for creating rehabilitation strategies. Revealing the connection between posture and cognitive level will not only reveal the positive effect of postural correlation on cognitive skills, but will also guide the importance of posture assessment in individuals with cognitive disorders.

ELIGIBILITY:
Inclusion Criteria:

- Athletes in early adolescence who voluntarily agreed to participate in the study will be included.

Exclusion Criteria:

* Presence of neurological and/or orthopedic and/or psychopathological disease, Having a history of visual, mental or systematic disease,
* The athlete's medical history has a history of major injury and/or surgery related to the lower extremity and trunk,
* Acute or chronic pain complaints will be determined as exclusion criteria.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Athletes in early adolescence
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Evaluation of cognitive functions | 20 April 2023
  The Stroop Test TBAG Form consists of four white cards measuring 14.0 cm x 21.5 cm. On each card, there are 6 rows consisting of 4 items arranged randomly. These cards are the 'stimulus' items of the test and the subject has to react to these stimuli, in other words, to perform the 'tasks'. The scores of the test are obtained by scoring the sections separately. In the Turkish version of the test performed by Karakaş et al., it was reported that the completion times of each section could be used. In the first two sections, it is required to read the words on the cards, and in the last three sections, the colors of the words or shapes are named. A stopwatch is used to measure reaction times. Time scores of the test; It is determined as the time from giving the 'start' command until the last item of the card is read/sung.
Evaluation of posture | 20 April 2023
  For posture assessment, the form of Corbin et al. will be applied. Individuals from lateral (head forward tilt, rounded back, shoulder protraction, kyphosis, lordotic changes, abdominal drooping, genu recurvatum, anterior balance) and posteriorly (lateral tilt of the head, shoulder inequality, protrusion of the scapula, scoliosis symptoms, presence of gibosity, lateral curvature of the spine) , hip inequality), each of the postural parameters in the form is scored by the physiotherapist according to its severity (0=absent, 1=mildly severe, 2=moderately severe, 3=good-severe). Postural status is classified according to the total score, by summing the scores of each parameter according to the severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)